CLINICAL TRIAL: NCT06038890
Title: The Learning Curve of Transurethral Holmium Laser Enucleation of the Prostate, Multicenter Prospective Assessment Through a Novel Technique
Brief Title: The Learning Curve of Transurethral Holmium Laser Enucleation of the Prostate, Prospective Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Professor of Urology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Mans.9.2023
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Learning Curve; Laser; Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: A single cohort of consecutively performed cases in participating centers done by new learners using the assigned technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holmium laser enculeation of the prostate (Experimental): veil-sparing Holmium laser enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of the prostate using the veil-sparing technique

INTERVENTIONS:
Procedure: Holmium laser enucleation of the prostate using the veil-sparing technique — Holmium laser enucleation of the prostate using the veil-sparing technique

SUMMARY:
Despite the high-quality evidence supporting the safety and efficacy of Holmium laser enucleation of the prostate (HOLEP), wide adoption of the procedure is hindered by learning difficulties. Veil-sparing HOLEP was popularized with a standardized approach to learning.

Prospective multicenter assessment of the learning curve of HoLEP through a novel technique with structured learning protocol.

Learning outcome measures will be assessed against time and number of performed cases of new learners in a multicenter study.

DETAILED DESCRIPTION:
INTRODUCTION Holmium laser enucleation of the prostate (HoLEP) was described in 1998 1 and since then, it has the highest level of evidence supporting its safety, efficacy and durability in treating benign prostate hyperplasia (BPH) 2.

Furthermore, it is a cost-effective alternative both in developing3 and developed4 countries. Nevertheless, learning difficulties hinder wide adoption of this technique among urologists and even more some centers discontinue doing this technique due complications encountered early in the learning curve5.

Performance of a task repetitively changes with experience over time. Plotting performance (outcome measures) against experience (number of performed tasks) produces a learning curve.

Improvement tends to be rapid at first and then tails off over time until a steady state is reached (Plateau) 6. Time-To-Plateau (TTP); number of HoLEP tasks is variably reported; 20-307-9, 5010 or even more procedures were reported as time needed to reach steady state (plateauing).

Elshal et al in 2023 compared this novel veil sparing approach in a comparitve study with the standard HOLEP approach and concluded that the veil sparing approach was associated with better short term urine continence.11 In this work we aim at assessment of the learning curve using this novel technique (Veil sparing HOLEP).

In this study, this novel technique is proposed to shorten the time to plateau (steady state) in mainly safety and efficiency outcome measures of HOLEP.

RATIONAL

Despite the high-quality evidence supporting the safety and efficacy of HOLEP, wide adoption of the procedure is hindered by learning difficulties. Veil-sparing HOLEP was popularized with a standardized approach for learning.

RESEARCH QUESTION Will Veil sparing Holmium laser enucleation with its standardized approach to learning cut short the learning curve?

HYPOTHESIS Veil-sparing Holmium laser enucleation of the prostate is feasible, and efficient, with a shorter learning curve.

AIM OF THE WORK We aim at assessment of the learning curve using this novel technique (Veil sparing HOLEP) In this study, this novel technique is proposed to shorten the time to plateau (steady state) in mainly safety and efficiency outcome measures of HOLEP.

PATIENTS AND METHODS

A. Study design:

Design: A Prospective multicenter cohort study. Sample size: Assuming that all cases met the inclusion and exclusion criteria will be included. During the study period (12 months), 4 cases/ month.48 cases will be included as a comprehensive sample.

Study population: eligible patients from our outpatient clinic, who are indicated for transurethral surgery for BPO will be screened for inclusion and exclusion criteria and will be offered informed consent.

B. Procedure:

1. Preoperative evaluation

   All patients will be subjected to:

   Written informed consent will be obtained from all patients Clinical history taking including International prostate symptom score (IPSS) and Quality of life (QoL).

   Physical and clinical examination Transrectal ultrasound (TRUS) to assess the prostate volume. PVRU by Pelvi-abdominal U/S (PA us). Uroflowmetry. Urine culture. Pre-operative routine laboratory investigations including CBC, PT, PTT, INR, liver and kidney functions.
2. Set-up Endoscopy: At our institution, we use a 26 French (Fr) continuous flow resectoscope with a laser bridge adapter and an endoscopic camera. The laser bridge adapter stabilizes the laser fiber and fixes it at the 6'oclock position on the endoscope. This set up helps keep the laser fiber at a fixed length from the tip of the endoscope and stabilizes the laser fiber.

   Laser machine: we use a 100-Watt holmium laser and an end-firing 550-micron laser fiber with energy settings of 2.0 J and frequency settings of 50 Hz.

   For tissue morcellation, a 26 Fr offset nephroscope is used along with a transurethral soft-tissue morcellator. The morcellator consists of two 5 mm reciprocating hollow metal blades, a hand-piece, a two-phase foot pedal, and a control box. The control box consists of a motor unit that powers the blades and supplies suction for tissue removal. A tissue collection device collects the chips as they are suctioned out of the bladder.
3. Points of the HOLEP technique Veil sparring HOLEP was performed in stepwise approach abbreviated for sake of learning as (IT PAS ABCD).11 Inspection of the prostate morphology looking for the main landmarks including the verumontanum, apical bulge, bladder neck and the ureteral orifices.

Incision of the prostate from the bladder neck to the verumontanum. The principle of the incision is to touch with the laser fiber and keep pressing the prostatic tissue using the scope.

Trough creation: the idea of trough creation is to create a working channel wider between the bladder neck and the verumontanum by hugging and pressing against the lateral lobes and trying to incise underneath each of them Plain development: the Incision is extended lateral to the verumontanum just mucosal incision following the apical bulge. Once the mucosal incision is completed, the laser fiber is withdrawn and using the tip of the scope bluntly enucleating the lateral lobes developing a plain between the surgical capsule and the prostatic adenoma.

Apico-lateral dissection: at this step the scope will be rotated 180 degrees where the laser fiber will come at 12 o'clock position, then compound sharp and blunt dissection of the prostatic adenoma from the prostatic surgical capsule progressing laterally trying to insinuate the scope between the surgical capsule and the prostatic adenoma.

Sphincter liberation (strip cutting): at this step, the scope will be gradually withdrawn out of the prostatic fossa looking for the sphincteric ring. Once the sphincteric ring is identified, we move the scope proximal to the ring to start cutting from 12 o'clock position towards the plain we previously created. We keep cutting only the mucosa we keep hugging the adenoma pressing on it trying to leave the veil of mucosa covering the sphincter ring.

Anterior dissection and commissurotomy: in this step we aim at creating an anterior plain connecting the laterally created plain to the anterior commissure. So, we keep curving anterior to the adenoma till we start anterior commissurotomy. Once the scope is riding the adenoma, we progress to the bladder neck connecting the lateral created plain to the anterior commissure cutting and sharply dissecting all residual attachment of the prostatic adenoma to the surgical capsule.

Bladder neck dissection: we start bladder neck dissection at 12 o'clock position where we start cutting anterior to the adenoma from the 12 o'clock position progressing laterally till 10 o'clock position.

C-shaped baso-lateral dissection: in this step we start sharp dissection cutting all around the adenoma in a c-shaped fashion progressively from the 10 o'clock position on the right lateral lobe towards the 7 o'clock position. This step entails circumferential dissection of the bladder neck fibers. The end of the c-shaped baso-lateral dissection is the identification of the ureteral orifices.

Detachment of the adenoma after its flipping inside the bladder: in this step we keep pressing the adenoma from underneath and lateral towards the bladder neck till the adenoma is flipped inside the bladder. Once the adenoma is flipped inside the bladder it will stretch its basal attachment so it is easier to be cut using the laser fiber from lateral to medial.

The other prostatic lobe will be enucleated in a similar way starting by Incision in front of the verumontanum with extension of the Incision following the apical bulge and later blunt enucleation.

The procedure will be concluded by tissue morcellation with extraction of the enucleated prostatic tissue.

Lastly carful inspection of the prostatic fossa, sphincteric ring covered by mucosal veil all around and anterior. Careful hemostasis will be done before ending the procedure.

Hemostasis is very good with this technique; however persistent small bleeders should be coagulated prior to morcellation. Coagulation is accomplished by defocusing the laser energy off any bleeding tissue. The desired result is that the tissue will blanch and stop bleeding.

Tissue morcellation The first step in tissue morcellation is to ensure the bladder is full. A 26 Fr offset nephroscope with the soft-tissue morcellator is inserted into the bladder. The blades of the morcellator should be placed in the center of the bladder away from the bladder mucosa. The two-phase foot pedal is then depressed to engage the suction but not the reciprocating blades. Adenoma is then drawn to the tip of morcellator blades. If the suction necessary to engage the adenoma will collapse the bladder too quickly, a second inflow tubing can be attached to the nephroscope outflow channel to increase the inflow and keep the bladder distended. Once the adenoma is at the tip of the morcellator, the foot pedal is depressed further, activating the blades, and the adenoma is morcellated, cutting the adenoma into small pieces that are suctioned out of the bladder and deposited in the collection chamber. Small pieces of the adenoma should not be chased with the morcellator blades in the bladder because of the increased risk of bladder injury.

Instead, the small adenomatous tissue should be removed by either a modified resectoscope loop, a rigid grasper for the nephroscope, Ellik evacuator or glass Toomey syringe. Once all chips are removed a 24 Fr three-way Foley catheter is inserted and bladder irrigation is instituted if needed.

Postoperative care If continuous bladder irrigation is used then usually it is continued only overnight. In the am of postoperative day 1 the bladder irrigation is discontinued once the hematuria stopped, and patients are given a trial of void. If they fail the trial of void, they are discharged home on postoperative day 1 with an 18 Fr Coude catheter for 3-5 days.

Follow-up assessment included CBC for Hb loss immediately postoperatively. Urine analysis (± culture if indicated), IPSS, QoL, Qmax and PVRU assessment after 1, 4 and 12 months post-operatively. PSA level will be tested at 4 months and then annually unless otherwise indicated.

In each visit, patients were verbally interrogated if they experience any episodes of urine incontinence (UI) and its associated condition as coughing or with certain movements; (SUI) stress urine incontinence, urgency; (UUI) urge urine incontinence or mixed UI. Any patient reported prolonged UI to 4 months or persistent at 12 months, was examined by standardized one-hour pad test. Grade of UI was objectively reported as grade (zero-4)12.

Outcome measures:

A) Operative efficacy measures include; enucleation efficiency (retrieved prostate tissue weight divided by enucleation time), operative efficiency (retrieved prostate tissue weight divided by total operative time) and laser to prostate ratio (L/P ratio; amount of consumed laser energy divided by retrieved prostate tissue weight).

B) Postoperative efficacy measures include; percent reduction of postoperative PSA. Median value of PSA levels at 4 and 12 months was used as postoperative PSA. Percent reduction was used as a surrogate marker of postoperative reduction in prostate volume.

C) Operative safety measures include; capsule violation, bladder wall injury (superficial or deep) and intraoperative bleeding necessitating blood transfusion or conversion to TURP. Moreover, perioperative hemoglobin and hematocrit value deficit (preoperative minus immediate postoperative value) were depicted.

D) Catheter duration, hospital stay and postoperative safety measures include 30-days postoperative complications.

E) Urinary flow outcome measures include IPSS, QOL (quality of life), Qmax (Peak flow rate) and PVR.

F) Urinary continence status at each follow-up visits using ICIQ-UI-SF Questionnaire and one hour pad test.

G) Need for reoperation for recurrent infravesical obstruction will be depicted.

1. Fraundorfer, M. R., Gilling, P. J.: Holmium: YAG laser enucleation of the prostate combined with mechanical morcellation: preliminary results. Eur Urol, 33: 69, 1998
2. Cornu, J. N., Ahyai, S., Bachmann, A. et al.: A Systematic Review and Meta- analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update Eur Urol, 2014
3. Elshal, A. M., Mekkawy, R., Laymon, M. et al.: Holmium laser enucleation of the prostate for treatment for large-sized benign prostate hyperplasia; is it a realistic endourologic alternative in developing country? World J Urol, 2015
4. Salonia, A., Suardi, N., Naspro, R. et al.: Holmium laser enucleation versus open prostatectomy for benign prostatic hyperplasia: an inpatient cost analysis. Urology, 68: 302, 2006
5. Robert, G., Cornu, J. N., Fourmarier, M. et al.: Multicenter prospective evaluation of the learning curve of holmium laser enucleation of the prostate (HoLEP). BJU Int, 2015
6. Hopper, A. N., Jamison, M. H., Lewis, W. G.: Learning curves in surgical practice. Postgrad Med J, 83: 777, 2007
7. Elzayat, E. A., Elhilali, M. M.: Holmium laser enucleation of the prostate (HoLEP): long-term results, reoperation rate, and possible impact of the learning curve. Eur Urol, 52: 1465, 2007
8. Du, C., Jin, X., Bai, F. et al.: Holmium laser enucleation of the prostate: the safety, efficacy, and learning experience in China. J Endourol, 22: 1031, 2008
9. Bae, J., Oh, S. J., Paick, J. S.: The learning curve for holmium laser enucleation of the prostate: a single-center experience. Korean J Urol, 51: 688, 2010
10. Shah, H. N., Mahajan, A. P., Sodha, H. S. et al.: Prospective evaluation of the learning curve for holmium laser enucleation of the prostate. J Urol, 177: 1468, 2007.
11. Ahmed Elshal, Mostafa Ghazy, Mahmoud Laymon, Fady Kamal V07-03 VEIL SPARRING HOLMIUM LASER ENUCLEATION OF THE PROSTATE; TECHNICAL EVOLUTION AND PRELIMINARY RESULTS OF RANDOMIZED TRIAL, Journal of Urology: April 2023 - Volume 209 - Issue Supplement 4 doi: 10.1097/JU.0000000000003288.03
12. Abrams, P., Cardozo, L., Fall, M. et al.: The standardization of terminology in lower urinary tract function: report from the standardization sub-committee of the International Continence Society. Urology, 61: 37, 2003.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate volume (≥40 cc) who are indicated for transurethral surgery for the BPO.

Exclusion Criteria:

* Patients with IPSS <13.
* Patients with Qmax >15 mL/s.
* Presence of urethral stricture.
* Patients with neurogenic bladder.
* Patients with prostate cancer.
* Patients with previous prostate surgery.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate surgery offered only for men
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
time to plateau in enucleation effeminacy | one year
  time needed to reach a fixed rate of grams of prostate tissue removed per unit time (minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided